CLINICAL TRIAL: NCT02080221
Title: BrUOG 292: FOLFOX-A For Metastatic Pancreatic Cancer: A Phase II Brown University Oncology Research Group Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Lifespan (Other); SouthCoast Medical Group (Other); Memorial hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 292
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: metastatic pancreatic cancer; pancreatic cancer; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOXA (Experimental): 1 cycle = 14 days Abraxane ®: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.
  Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)
  Interventions: Drug: FOLFOXA

INTERVENTIONS:
Drug: FOLFOXA
  Other Names: 1 cycle = 14 days; Abraxane ®: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.; Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days; Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days; 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)

SUMMARY:
A standard treatment for your cancer is called FOLFIRINOX (this utilizes the FDA approved chemotherapy drugs fluorouracil, leucovorin, oxaliplatin and irinotecan). In this study you will receive the chemotherapy treatment FOLFOX-A (fluorouracil, oxaliplatin, leucovorin and Abraxane ®) which substitutes irinotecan for the FDA approved chemotherapy drug Abraxane ®. Even though Abraxane is FDA approved for pancreatic cancer, the combination of Abraxane with the other 3 drugs is being investigated. Your doctors are studying the activity and side effects of FOLFOX-A in advanced (metastatic) pancreatic cancer.

DETAILED DESCRIPTION:
See summary above

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytological confirmed pancreatic ductal adenocarcinoma. Patients with pathology or cytology showing carcinoma of pancreas or adenosquamous of the pancreas are also eligible.
2. Metastatic advanced disease.
3. No prior chemotherapy for pancreatic cancer
4. No major surgery within 3 weeks of the start of study treatment. Patients must have recovered from the side effects of any major surgery at the start of study treatment. For questions on if a surgery is deemed "major," definition by surgeon can be used for clarification. Laparoscopy and central venous catheter placement are not considered major surgery.
5. No prior invasive malignancy within the prior two years. However, patients with an early stage malignancy that is not expected to require treatment in the next 2 years (such as early stage, resected breast cancer or asymptomatic prostate cancer) are eligible.
6. ECOG performance status 0 or 1.
7. Age ≥ 18
8. Not pregnant and not nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to beginning of treatment. Post-menopausal women (surgical menopause or lack of menses >12 months) do not need to have a pregnancy test, please document status.
9. Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment. Documentation of this being discussed required.
10. Required Initial Laboratory Values:

    * Neutrophils ≥ 1,500/mm3
    * Platelet count ≥ 100,000/mm3
    * Creatinine ≤ 1.5 mg/dL -or- creatinine clearance ≥ 60 mL/min
    * Total bilirubin ≤ 1.25 x ULN
    * AST (SGOT) & ALT (SGPT) ≤ 2.5 x ULN (for patients with liver metastases, AST&ALT < 5xULN)
    * Alkaline phosphatase < 2.5xULN, unless bone metastasis is present and in the absence of liver metastasis

Exclusion Criteria:

1. Patients with known brain metastases
2. Prior hypersensitivity to Oxaliplatin or Abraxane ® that in the investigators opinion would put the patient at risk if re-exposed
3. Preexisting neuropathy
4. Patients with serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive FOLFOX-A 5. Patients with unstable biliary stents or with plastic stents. Information on type of stent is required at registration.

6. Patients with active infection or fever (patients on antibiotics for infection or patients getting over a cold or seasonal virus are not excluded), or known historical or active infection with HIV, hepatitis B, or hepatitis C.

7. Patients with sepsis or pneumonitis. 8. Patients with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies that in the investigator's opinion would put the patient at an increased risk.

10. Uncontrolled diabetes. If patient has diabetes, confirmation on status (controlled or uncontrolled) required at registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2020-01-09 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — BrUOG
Locations (2):
- United States (2):
  - Southcoast centers for cancer care, Fairhaven, Massachusetts
  - Lifespan Hospitals (The Miriam and RI Hospital, East Greenwich, Newport), Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOXA: 1 cycle = 14 days Abraxane ®: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.
  Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)
  FOLFOXA
Period: Overall Study
Arm/Group | FOLFOXA
Started | 50
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Clinical Progression of Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOXA
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 32
Age, Continuous [Mean (Full Range); unit: years] | 66 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 46
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Survival for Patients With Metastatic Pancreatic Cancer With First-line Treatment With FOLFOX-A as Compared to Historical Controls of Gemcitabine Alone.
Time Frame: Every 3 months for up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOXA
Number analyzed (Participants) | 48
months
  Progression- free survival | 5 [3 to 7]
  Overall survival | 11 [8 to 14]

2. Secondary Outcome: Response of Patients With Metastatic Pancreatic Cancer Who Receive the FOLFOX-A Regimen
Time Frame: Every 3 months for up to 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOXA
Number analyzed (Participants) | 48
Participants
  Complete response | 2
  Partial response | 12
  Stable disease | 12
  Progressive disease | 22

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | FOLFOXA
All-Cause Mortality (participants affected / at risk) | 2/48
Serious Adverse Events (participants affected / at risk) | 10/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXA (N=48)
Hyperglycemia (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hemoptysis (Blood and lymphatic system disorders) | 1
Acidosis (Blood and lymphatic system disorders) | 1
Acute kidney injury (Injury, poisoning and procedural complications) | 2
Anemia (Blood and lymphatic system disorders) | 1
Infection (Infections and infestations) | 5
Constipation (Gastrointestinal disorders) | 1
Lethargy (Nervous system disorders) | 1
Multi organ failure (General disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pain (General disorders) | 4
Peritonitis (Infections and infestations) | 1
Thrombocytopenia (Investigations) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Small bowel obstruction (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Stroke (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Blood bilirubin elevated (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 5
Sepsis (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXA (N=48)
Neutropenia (Investigations) | 21
Thrombocytopenia (Investigations) | 36
Anemia (Blood and lymphatic system disorders) | 30
Peripheral sensory neuropathy (Nervous system disorders) | 33
Diarrhea (Gastrointestinal disorders) | 20
Anorexia (Metabolism and nutrition disorders) | 13
Vomiting (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 36
Mucositis oral (Gastrointestinal disorders) | 6
Arthralgia (Nervous system disorders) | 2
Weight loss (Investigations) | 30
Elevated AST/ALT (Investigations) | 22
Elevated alkaline phosphatase (Investigations) | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT02080221/Prot_SAP_ICF_000.pdf